CLINICAL TRIAL: NCT03365791
Title: Modular Phase 2 Study to Link Combination Immune-therapy to Patients With Advanced Solid and Hematologic Malignancies. Module 9: PDR001 Plus LAG525 for Patients With Advanced Solid and Hematologic Malignancies.
Brief Title: PDR001 Plus LAG525 for Patients With Advanced Solid and Hematologic Malignancies
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CPDR001XUS01
Record Dates: First submitted 2017-11-20; First posted 2017-12-07 (Actual); Results first posted 2021-04-19 (Actual); Last update posted 2022-05-27 (Actual); Status verified 2022-05

CONDITIONS: Small Cell Lung Cancer; Gastric Adenocarcinoma; Esophageal Adenocarcinoma; Castration Resistant Prostate Adenocarcinoma; Soft Tissue Sarcoma; Ovarian Adenocarcinoma; Advanced Well-differentiated Neuroendocrine Tumors; Diffuse Large B Cell Lymphoma
Keywords: PDR001; LAG525; Immune checkpoint blockade; Solid tumor malignancy; lymphoma; Small cell lung cancer (SCLC); Gastric/esophageal adenocarcinoma; Castration resistant prostate adenocarcinoma (CRPC); Soft tissue sarcoma; Ovarian adenocarcinoma; Advanced well-differentiated neuroendocrine tumors (NETs); Diffuse large B cell lymphoma (DLBCL)
MeSH Terms: conditions — Small Cell Lung Carcinoma; Adenocarcinoma Of Esophagus; Sarcoma; Lymphoma, Large B-Cell, Diffuse; Lymphoma | interventions — spartalizumab

STUDY DESIGN:
Intervention Model Description: This is a phase II, open-label, study to determine the efficacy and safety of treatment with the combination of PDR001+LAG525 across multiple tumor types that are relapsed and/or refractory to available standard of care therapies. Patients will receive study treatment for a maximum of 2 years. All disease assessments will be performed locally by the investigator.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- PDR001+LAG525 (Experimental): PDR001 300 mg and LAG525 400 mg administered via i.v. infusion over 30 minutes once every 3 weeks (Q3W). LAG525 was given first followed by PDR001.
  Interventions: Biological: PDR001; Biological: LAG525

INTERVENTIONS:
Biological: PDR001 — PDR001 is a high-affinity, ligand-blocking, humanized anti-programmed death-1 (PD-1) IgG4 antibody that blocks the binding of Programmed death-ligand 1 (PD-L1) and programmed death-ligand 2 (PD-L2) to PD-1.
Biological: LAG525 — LAG525 is a high-affinity, ligand-blocking, humanized anti-LAG-3 IgG4 antibody which blocks the binding of the known LAG-3 ligand MHC class II to LAG-3.

SUMMARY:
The purpose of this signal seeking study is to determine whether treatment with PDR001 and LAG525 demonstrates sufficient efficacy in advanced malignancies to warrant further study.

DETAILED DESCRIPTION:
This was a phase II, open-label study to determine the efficacy and safety of treatment with the combination of PDR001+LAG525 across multiple tumor types that are relapsed and/or refractory to available standard of care therapies. There were 7 tumor cohorts assessed: 1) Small cell lung cancer, 2) Gastric/esophageal adenocarcinoma, 3) Castration resistant prostate adenocarcinoma (CRPC), 4) Soft tissue sarcoma, 5) Ovarian adenocarcinoma, 6) Advanced well-differentiated neuroendocrine tumors and 7) Diffuse large B cell lymphoma (DLBCL).

Participants were treated with the combination of PDR001 300 mg with LAG525 400 mg once every 3 weeks (Q3W) via intravenous (i.v.) infusion. Participants received study treatment for a maximum of 2 years, or until disease progression (assessed by investigator per Response Evaluation Criteria In Solid Tumors version 1.1 (RECIST 1.1) or the Revised Response Criteria for Malignant Lymphoma criteria (Cheson et al 2007)), unacceptable toxicity, death or discontinuation from study treatment for any other reason.

ELIGIBILITY:
Inclusion Criteria:

Patients eligible for inclusion in this study had to meet all of the following criteria:

* Patient must have had at least one prior line of therapy for their disease and must not be beyond 4th progression/relapse of disease (5 maximum prior lines).
* Patient has a pathology confirmed diagnosis of a solid tumor or lymphoma listed in the section "condition". Patients must have measurable disease as per appropriate guidelines (Solid Tumors by RECIST 1.1 and Diffuse Large B-cell Lymphoma by Revised Response Criteria for Malignant Lymphoma - Cheson et al 2007).

Exclusion Criteria:

Patients eligible for this study must not meet any of the following criteria:

* History of severe hypersensitivity reactions to other monoclonal antibodies.
* Impaired cardiac function or clinically significant cardiac disease.
* Active, known or suspected autoimmune disease or a documented history of autoimmune disease within three years prior to screening with a few exceptions as per protocol.
* Patients previously exposed to anti-PD-1/PD-L1 treatment who are adequately treated for skin rash or with replacement therapy for endocrinopathies should not be excluded.
* Patient with second primary malignancy within < 3 years of first dose of study treatment.
* Prior immunotherapy treatment with PD-1, PD-L1, CTLA-4, or LAG-3 antibodies.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2018-01-24 (Actual); Primary Completion 2019-02-21 (Actual); Study Completion 2020-09-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (20):
- United States (20):
  - California Pacific Medical Center Drug Shipment (2), San Francisco, California
  - Hematology Oncology Associates of the Treasure Coast, Port Saint Lucie, Florida
  - University Cancer and Blood Center, LLC, Athens, Georgia
  - Northwestern University Medical School, Chicago, Illinois
  - University of Illinois Cancer Center at Chicago SC, Chicago, Illinois
  - Illinois Cancer Care P.C. Jesse Brown VA, Peoria, Illinois
  - Indiana University, Indianapolis, Indiana
  - University of Iowa Hospitals and Clinics Comprehensive Cancer Center, Iowa City, Iowa
  - The University of Kansas Clinical Research Center, Fairway, Kansas
  - Weinberg Cancer Institute at Franklin Square Hospital, Baltimore, Maryland
  - Billings Clinic Dept of Billings Clinic(2), Billings, Montana
  - Oncology Hematology West Nebraska Cancer Specialists, Omaha, Nebraska
  - Comprehensive Cancer Centers, Las Vegas, Nevada
  - Oregon Health and Science University, Portland, Oregon
  - Oncology Consultants Oncology Consultants, Houston, Texas
  - University of Texas - MD Anderson Cancer Center, Houston, Texas
  - Kadlec Clinic Hematology and Oncology, Kennewick, Washington
  - Providence Regional Cancer System SC, Lacey, Washington
  - University of Wisconsin Hospital and Clinics, Madison, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations. This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com.

REFERENCES:
- See also: A Plain Language Trial Summary is available on novctrd.com — https://www.novctrd.com/ctrdweb/patientsummary/patientsummaries?patientSummaryId=974

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in 20 investigative sites in 1 country (United States).
Pre-assignment Details: The screening period began once patients had signed the study informed consent. All screening evaluations were performed as closely as possible to the beginning of treatment and never more than 21 days prior to starting study treatment. After screening, the treatment period started on Cycle 1 Day 1.
Period: Overall Study
Arm/Group | PDR001+LAG525
Started | 76
Full Analysis Set (FAS) (The FAS includes all participants who received at least one dose of study treatment and had at least one valid post-baseline efficacy assessment.) | 75
Completed | 4
Not Completed | 72
Not completed — Adverse Event | 5
Not completed — Death | 1
Not completed — Lost to Follow-up | 1
Not completed — Physician Decision | 9
Not completed — Progressive disease | 51
Not completed — Subject/guardian decision | 5

BASELINE CHARACTERISTICS:
Arm/Group | PDR001+LAG525
Number analyzed (Participants) | 76
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.1 (10.57)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31
  Male | 45
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 1
  Black | 1
  Caucasian | 67
  Unknown | 7

OUTCOME MEASURES:

1. Primary Outcome: Clinical Benefit Rate (CBR) at 24 Weeks of PDR001+LAG525 by Tumor Type in Multiple Solid Tumors and Lymphoma
Description: CBR is defined as the percentage of participants with a best overall response of Complete Response (CR), Partial Response (PR) and Stable Disease (SD). Tumor response was based on local investigator assessment. For participants with solid tumors the assessment criteria was Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST v1.1) and for participants with lymphoma the assessment criteria was the Revised Response Criteria for Malignant Lymphoma (Cheson et al 2007).
  For RECIST v1.1, CR=Disappearance of all non-nodal target lesions. In addition, any pathological lymph nodes assigned as target lesions must have a reduction in short axis to < 10 mm; PR= At least a 30% decrease in the sum of diameter of all target lesions, taking as reference the baseline sum of diameters; SD= Neither sufficient shrinkage to qualify for PR or CR nor an increase in lesions which would qualify for progression.
  CBR (CR+PR+SD) is reported overall and by tumor type.
Time Frame: 24 weeks
Population: Full Analysis Set (FAS)
Measure: Count of Participants; unit: Participants
Arm/Group | PDR001+LAG525
Number analyzed (Participants) | 75
Participants
  Overall | 25
  Small cell lung cancer: number analyzed (Participants) | 16
  Small cell lung cancer | 3
  Gastric/esophageal adenocarcinoma: number analyzed (Participants) | 13
  Gastric/esophageal adenocarcinoma | 2
  Castration resistant prostate adenocarcinoma (CRPC): number analyzed (Participants) | 10
  Castration resistant prostate adenocarcinoma (CRPC) | 5
  Soft tissue sarcoma: number analyzed (Participants) | 10
  Soft tissue sarcoma | 4
  Ovarian adenocarcinoma: number analyzed (Participants) | 10
  Ovarian adenocarcinoma | 2
  Advanced well-differentiated neuroendocrine tumors: number analyzed (Participants) | 7
  Advanced well-differentiated neuroendocrine tumors | 6
  Diffuse large B cell lymphoma (DLBCL): number analyzed (Participants) | 9
  Diffuse large B cell lymphoma (DLBCL) | 3

2. Secondary Outcome: Overall Response Rate (ORR)
Description: ORR is defined as the percentage of participants with a best overall response of Complete Response (CR) or Partial Response (PR). Tumor response was based on local investigator assessment. For participants with solid tumors the assessment criteria was Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST v1.1) and for participants with lymphoma the assessment criteria was the Revised Response Criteria for Malignant Lymphoma (Cheson et al 2007).
  For RECIST v1.1, CR=Disappearance of all non-nodal target lesions. In addition, any pathological lymph nodes assigned as target lesions must have a reduction in short axis to < 10 mm; PR= At least a 30% decrease in the sum of diameter of all target lesions, taking as reference the baseline sum of diameters.
  ORR (CR+PR) is reported overall (including all tumor types).
Time Frame: From start of treatment until end of treatment, assessed up to 113 weeks
Population: Full Analysis Set (FAS)
Measure: Count of Participants; unit: Participants
Arm/Group | PDR001+LAG525
Number analyzed (Participants) | 75
Participants | 7

3. Secondary Outcome: Time to Response (TTR)
Description: TTR is defined as the time from the date of first dose to the date of first documented response of Complete Response (CR) or Partial Response (PR). In case of solid tumor if a patient did not achieve a confirmed response they were censored at maximum follow-up for patients who had a PFS event (progressed or died due to any cause), or at last adequate tumor assessment date otherwise.
  Tumor response was based on local investigator assessment. For participants with solid tumors the assessment criteria was Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST v1.1) and for participants with lymphoma the assessment criteria was the Revised Response Criteria for Malignant Lymphoma (Cheson et al 2007).
Time Frame: From start of treatment to the first documented response of either complete response or partial response, assessed up to 113 weeks
Population: Full Analysis Set (FAS)
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | PDR001+LAG525
Number analyzed (Participants) | 75
months | NA [NA to NA] — Not estimable due to insufficient number of participants with events.

4. Secondary Outcome: Duration of Response (DOR)
Description: DOR only applies to subjects for whom best overall response is complete response (CR) or partial response (PR). DOR is defined as the time between the date of first documented response (CR or PR) and the date of first documented progression/relapse or death due to any cause within 150 days of the last study drug dose date. If a patient not had an event, duration was censored at the date of last adequate tumor assessment.
  Tumor response was based on local investigator assessment. For participants with solid tumors the assessment criteria was Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST v1.1) and for participants with lymphoma the assessment criteria was the Revised Response Criteria for Malignant Lymphoma (Cheson et al 2007).
Time Frame: From first documented response (CR or PR) to first documented progression or death, assessed up to 113 weeks
Population: Participants in the Full Analysis Set (FAS) for whom best overall response is complete response (CR) or partial response (PR)
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | PDR001+LAG525
Number analyzed (Participants) | 7
months | NA [5.8 to NA] — Not estimable due to insufficient number of participants with events.

5. Secondary Outcome: Time to Progression (TTP)
Description: TTP is the time from start of treatment to the date of event defined as the first documented progression or death due to underlying cancer. If a patient not had an event, time to progression was censored at the date of last adequate tumor assessment.
  Tumor response was based on local investigator assessment. For participants with solid tumors the assessment criteria was Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST v1.1) and for participants with lymphoma the assessment criteria was the Revised Response Criteria for Malignant Lymphoma (Cheson et al 2007).
Time Frame: From start of treatment to first documented progression or death due to underlying cancer, assessed up to 113 weeks
Population: Full Analysis Set (FAS)
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | PDR001+LAG525
Number analyzed (Participants) | 75
months | 2.8 [2.7 to 3.8]

6. Secondary Outcome: Progression-Free Survival (PFS)
Description: PFS is the time from the date of start of treatment to the date of event defined as the first documented progression or death due to any cause within 150 days of the last dose. If a patient has not had an event, progression-free survival is censored at the date of last adequate tumor assessment.
  Tumor response was based on local investigator assessment. For participants with solid tumors the assessment criteria was Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST v1.1) and for participants with lymphoma the assessment criteria was the Revised Response Criteria for Malignant Lymphoma (Cheson et al 2007).
Time Frame: From start of treatment to first documented progression or death, assessed up to 113 weeks
Population: Full Analysis Set (FAS)
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | PDR001+LAG525
Number analyzed (Participants) | 75
months | 2.8 [2.6 to 3.1]

7. Secondary Outcome: Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: Number of participants with AEs and SAEs including changes in laboratory parameters, vital signs and ECGs qualifying and reported as AEs.
Time Frame: From first dose of study treatment until last dose of study treatment plus 150 days post treatment, assessed up to 135 weeks.
Population: All participants who received at least one dose of study treatment
Measure: Count of Participants; unit: Participants
Arm/Group | PDR001+LAG525
Number analyzed (Participants) | 76
Participants
  AEs | 75
  SAEs | 32

8. Secondary Outcome: Number of Participants With Dose Interruptions and Permanent Discontinuation of Study Drug
Description: Number of participants with at least one dose interruption of PDR001 and LAG525 and number of participants with permanent dose discontinuation of PDR001 and LAG525.
Time Frame: From first dose of study treatment until last dose of study treatment, assessed up to 113 weeks.
Population: All participants who received at least one dose of study treatment
Measure: Count of Participants; unit: Participants
Arm/Group | PDR001+LAG525
Number analyzed (Participants) | 76
Participants
  PDR001 - dose interruption | 30
  PDR001 - permanent dose discontinuation | 72
  LAG525 - dose interruption | 30
  LAG525 - permanent dose discontinuation | 72

9. Secondary Outcome: Dose Intensity
Description: Dose intensity (mg/day) of PDR001 and LAG525 is calculated as cumulative dose in milligrams divided by duration of exposure in days.
Time Frame: From first dose of study treatment until last dose of study treatment, assessed up to 113 weeks.
Population: All participants who received at least one dose of study treatment
Measure: Mean (Standard Deviation); unit: mg/day
Arm/Group | PDR001+LAG525
Number analyzed (Participants) | 76
mg/day
  PDR001 | 14.1 (0.88)
  LAG525 | 18.8 (1.20)

ADVERSE EVENTS:
Time Frame: In the on-treatment period, adverse events (AEs) and serious AEs (including the All-Cause Mortality data table) are presented from first dose of study treatment until last dose of study treatment plus 30 days post treatment. In the extended safety follow-up period, AEs and serious AEs (including the All-Cause Mortality data table) are presented from day 31 to day 150 after last administration of study treatment.
Description: In the on-treatment period, any sign or symptom that occurs during the study treatment plus 30 days post treatment.
  In the extended safety follow-up period, any sign or symptom that occurs between 31 and 150 days post treatment.
Groups:
- PDR001+LAG525 On-treatment Period; PDR001+LAG525 Extended Safety Follow-up Period: PDR001 300 mg and LAG525 400 mg administered via i.v. infusion over 30 minutes once every 3 weeks (Q3W). LAG525 was given first followed by PDR001
Arm/Group | PDR001+LAG525 On-treatment Period | PDR001+LAG525 Extended Safety Follow-up Period
All-Cause Mortality (participants affected / at risk) | 9/76 | 18/76
Serious Adverse Events (participants affected / at risk) | 31/76 | 4/76
Other Adverse Events (participants affected / at risk) | 74/76 | 12/76
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PDR001+LAG525 On-treatment Period (N=76) | PDR001+LAG525 Extended Safety Follow-up Period (N=76)
Lymphadenopathy (Blood and lymphatic system disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 0
Atrial flutter (Cardiac disorders) | 1 | 0
Cardiac failure congestive (Cardiac disorders) | 1 | 0
Pericardial effusion (Cardiac disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 2 | 0
Abdominal pain lower (Gastrointestinal disorders) | 1 | 0
Haematemesis (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 2 | 0
Vomiting (Gastrointestinal disorders) | 2 | 0
Asthenia (General disorders) | 3 | 0
Infusion related reaction (General disorders) | 1 | 0
Autoimmune hepatitis (Hepatobiliary disorders) | 1 | 0
Bacteraemia (Infections and infestations) | 1 | 0
Clostridium difficile infection (Infections and infestations) | 1 | 0
Enterocolitis infectious (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 5 | 0
Pyelonephritis (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0
Alanine aminotransferase increased (Investigations) | 1 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 0
Weight decreased (Investigations) | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Myelitis transverse (Nervous system disorders) | 1 | 1
Failure to thrive (Psychiatric disorders) | 1 | 0
Mental status changes (Psychiatric disorders) | 1 | 0
Haematuria (Renal and urinary disorders) | 1 | 0
Urinary retention (Renal and urinary disorders) | 1 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Superior vena cava syndrome (Vascular disorders) | 1 | 0
Ventricular extrasystoles (Cardiac disorders) | 0 | 1
Spinal cord compression (Nervous system disorders) | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | PDR001+LAG525 On-treatment Period (N=76) | PDR001+LAG525 Extended Safety Follow-up Period (N=76)
Anaemia (Blood and lymphatic system disorders) | 13 | 2
Dizziness (Cardiac disorders) | 6 | 2
Dyspnoea (Cardiac disorders) | 18 | 1
Oedema peripheral (Cardiac disorders) | 10 | 1
Hypercalcaemia (Endocrine disorders) | 5 | 0
Dry eye (Eye disorders) | 4 | 0
Abdominal distension (Gastrointestinal disorders) | 8 | 0
Abdominal pain (Gastrointestinal disorders) | 14 | 0
Constipation (Gastrointestinal disorders) | 20 | 0
Diarrhoea (Gastrointestinal disorders) | 15 | 1
Dry mouth (Gastrointestinal disorders) | 6 | 0
Dysgeusia (Gastrointestinal disorders) | 4 | 0
Dyspepsia (Gastrointestinal disorders) | 4 | 1
Dysphagia (Gastrointestinal disorders) | 4 | 0
Flatulence (Gastrointestinal disorders) | 5 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 4 | 0
Nausea (Gastrointestinal disorders) | 26 | 1
Vomiting (Gastrointestinal disorders) | 20 | 0
Chills (General disorders) | 6 | 0
Fatigue (General disorders) | 28 | 0
Non-cardiac chest pain (General disorders) | 4 | 0
Pyrexia (General disorders) | 7 | 0
Ascites (Hepatobiliary disorders) | 5 | 1
Urinary tract infection (Infections and infestations) | 4 | 1
Fall (Injury, poisoning and procedural complications) | 7 | 1
Aspartate aminotransferase increased (Investigations) | 5 | 0
Blood alkaline phosphatase increased (Investigations) | 5 | 0
Blood creatinine increased (Investigations) | 10 | 0
Weight decreased (Investigations) | 7 | 0
Decreased appetite (Metabolism and nutrition disorders) | 22 | 0
Dehydration (Metabolism and nutrition disorders) | 9 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 6 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 10 | 0
Hypothyroidism (Metabolism and nutrition disorders) | 6 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 7 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 13 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 7 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 4 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 8 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 4 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 | 0
Headache (Nervous system disorders) | 11 | 0
Insomnia (Nervous system disorders) | 8 | 1
Anxiety (Psychiatric disorders) | 6 | 0
Depression (Psychiatric disorders) | 6 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 12 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 5 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 6 | 1
Rash (Skin and subcutaneous tissue disorders) | 9 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 6 | 2
Hypertension (Vascular disorders) | 4 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. Novartis does not prohibit any investigator from publishing. Any publications from a single site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2018-07-16): https://cdn.clinicaltrials.gov/large-docs/91/NCT03365791/Prot_001.pdf
  • Statistical Analysis Plan (2021-02-03): https://cdn.clinicaltrials.gov/large-docs/91/NCT03365791/SAP_000.pdf